CLINICAL TRIAL: NCT06082804
Title: Evaluation of Advanced Practice Nurse's Management of Patients with Chronic Myeloid Leukemia
Acronym: IPA-LMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Duffaut - Avignon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPA-LMC
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Chronic Myelogenous Leukemia - Chronic Phase
Keywords: Advanced Practice Nursing; Quality of life; Adverse event
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Practice Management, Medical

STUDY DESIGN:
Intervention Model Description: 60 patients will be included, these patients will be randomized into two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: IPA group (Experimental): Patients in arm A are followed by the advanced practice nurse and the hematologist.
  Interventions: Other: APN and medical management; Behavioral: Quality of life assessment; Behavioral: Treatment compliance assessment
- B: Control group (Active Comparator): Patients in arm B are followed by the hematologist only (standard of care).
  Interventions: Other: Medical management; Behavioral: Quality of life assessment; Behavioral: Treatment compliance assessment

INTERVENTIONS:
Other: APN and medical management — Patients are followed by the advanced practice nurse and the hematologist.
  Arms: A: IPA group
Other: Medical management — Patients are followed by the hematologist only (standard of care).
  Arms: B: Control group
Behavioral: Quality of life assessment — EORTC-QLQ-C30 questionnaire
Behavioral: Treatment compliance assessment — GIRERD questionnaire

SUMMARY:
Chronic Myeloid Leukemia (CML) affects 820 people per year in France (2018), half of them are older than 60 years old.

Tyrosine Kinase Inhibitors (TKI) are new kind of targeted therapy whose efficiency allow for a high rate of complete molecular response, leading to a disruption of treatment under certain conditions.

Optimizing CML treatment is a major concern, particularly for adverse events management, treatment compliance and therapeutic response. Multiple studies demonstrated that grade ≤ II adverse events are most likely to be under reported by patients and clinicians. Although these adverse events are mostly reported by clinical examination, needing minimal treatment. These toxicities could alter daily and domestic living activities, potentially impacting treatment compliance and therapeutic response. Therefore, early detection of these adverse events is a major challenge for the prognosis and care of CML.

The Advanced Practice Nurse (APN), a new health care professional, acquired the skills needed to independently follow, manage and care the patients with medical approvals.

At international level, many studies, in oncology and in others domains, have been done to demonstrate the added value of the APN, particularly in improving patient's quality of life, management, care of drug-induced adverse events and treatment compliance.

In France, because of the recentness of the profession, only few studies were have been conducted. The goal of this study is to demonstrate the benefit of APN in clinical follow-up, quality of life, treatment compliance, and therapeutic response of CML patients. These effects could be managed thanks to early detection and management of ≤ grade II adverse events during consultation, in partnership with the patients, and in collaborative working.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* CML patient in chronic phase, eligible for oral therapy.
* Newly diagnosed CML and/or initiating oral therapy :

  * Patient changing treatment for non-response or loss of therapeutic response or toxicities, on the condition that these toxicities are resolved or grade I maximum at the time of inclusion.
  * Newly start of oral therapy.
* Patient eligible to a follow-up by an advanced practice nurse.
* Patient capable to understand french and complete a questionnaire.

Exclusion Criteria:

* Patient that had a follow-up > 3 months by an advanced practice nurse for CML before inclusion.
* Patient changing treatment for toxicities, if these toxicities are still > grade I at inclusion.
* Patient enrolled in another interventional research protocol for CML.
* Pregnant women.
* Patient under legal protection, deprived of liberty or unable to be included in a research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the role of the advanced practice nurse in early detection of grade I-II adverse events during care and management of Chronic Myeloid Leukemia compared to standard of care (hematologist only). | Inclusion and 6 months
  Grade I-II adverse events rate

SECONDARY OUTCOMES:
Evaluate the role of the advanced practice nurse in early detection of grade I-II adverse events during care and management of Chronic Myeloid Leukemia compared to standard of care (hematologist only). | 6 months and 12 months
  Grade I-II adverse events rate
Assessment of patient's quality of life | Inclusion, 6 months and 12 months
  European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 : EORTC-QLQ-C30 (composed of both multi-item scales and single-item measures : 5 functional scales, 3 symptom scales, 6 single items and a global health status. All of the the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. ie : A high score for a functional scale represents a high level of functioning, a high score for the global health status represents a high quality of life but a high score for a symptom scale or a single item represents a high level of symptomatology).
Assessment of patient's compliance to treatment | 6 months and 12 months
  GIRERD questionnaire (measures range from 0 to 6. A low score represents a high level of compliance).
Grade > II adverse events rates | 6 months and 12 months
Hospitalization rate | 6 months and 12 months
Treatment discontinuation rate and/or treatment change rate | Every medical consultation, from inclusion to 12 months
Consultation time comparison between advanced practice nurse and hematologist | Every medical consultation, from inclusion to 12 months
Molecular response rate assessment | 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Tosello, APN, Principal Investigator — Centre Hospitalier d'Avignon, Service d'Oncologie Médicale-Hématologie Clinique
Locations (1):
- Centre Hospitalier d'Avignon, Hôpital Henri Duffaut, Avignon, France